CLINICAL TRIAL: NCT07180771
Title: A Phase II, Single-arm, Multicenter, Open Label Study to Evaluate Efficacy and Safety of BR101801 Monotherapy in Relapsed/Refractory Peripheral T-cell Lymphoma Patients
Brief Title: A Study of Bosmolisib (BR101801) in Participants With R/R PTCL.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-101801-CT-201
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: PTCL; Bosmolisib; BR101801; PI3K inhibitor; DNA-PK
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR101801 (Bosmolisib) (Experimental): Patients will receive BR101801 capsules orally, QD in 28-day cycles
  Interventions: Drug: BR101801

INTERVENTIONS:
Drug: BR101801 — Patients will receive 200mg capsules (100mg+100mg)
  Other Names: Bosmolisib

SUMMARY:
The objective of this phase II study is to evaluate the efficacy and safety of BR101801 in patients with peripheral T-cell lymphoma(PTCL).

DETAILED DESCRIPTION:
This phase II study will evaluate the efficacy and safety of single-dose BR101801 once daily in patients with peripheral T-cell lymphoma.

ELIGIBILITY:
Key Inclusion Criteria:

1. The ECOG performance status ≤ 2.
2. Life expectancy more than 3 months.
3. Patients with relapsed and/or refractory to standard therapy or are intolerance to standard therapy diagnosed with 2022 World Health Organization (WHO) classification

   * Peripheral T-cell lymphoma, not otherwise specified
   * Nodal TFH cell lymphoma, angioimmunoblastic-type
   * Nodal TFH cell lymphoma, follicular-type
   * Nodal TFH cell lymphoma, NOS
4. Patients currently requiring systemic therapy at the investigator's discretion.
5. Patients with a lesion measuring 1.5 cm or more in its longest transverse diameter, as determined by CT, PET/CT or MRI scans according to the 2014 Lugano criteria.

Key Exclusion Criteria:

1. The presence of overt leptomeningeal or active central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy or increasing doses of corticosteroids within the prior 2 weeks.
2. Impaired cardiac function or clinically significant cardiac disease.
3. Patients with interstitial pneumonia or history of drug-induced interstitial pneumonia/pneumonitis.
4. For patients with lymphoma:

   * Systemic antineoplastic therapy (including cytotoxic chemotherapy, alfa-interferon [INF], and toxin immunoconjugates) or any experimental therapy within 3 weeks or 5 half lives, whichever is shorter, before the first dose of study treatment.
   * Therapy with tyrosine kinase inhibitor within 5 half-lives before the first dose of study treatment.
   * Unconjugated monoclonal antibody therapies < 6 weeks before the first dose of study treatment.
5. Patients receiving systemic chronic steroid therapy or any immunosuppressive therapy (>20 mg/day prednisone or equivalent).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) (CR + PR) assessed by a blinded independent reviewer at the central lab according to the 2014 Lugano criteria | Up to 2 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (CR + PR) assessed by a blinded independent reviewer at the central lab according to the 2014 Lugano criteria | Up to 2 years
Overall Survival (OS) | Up to 2 years
Disease Control Rate (DCR) | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Progression-free Survival (PFS) | Up to 2 years
Time to Tumor Progression (TTP) | Up to 2 years
Quality of life assessment Using the EQ-5D-5L assessment | Every 2 cycles for up to 24 months (each cycle is 28 days)
  European quality of life 5 dimensions questionnaire. The values is 0 to 1, whereby 0 indicates death and 1 perfect health
Quality of life assessment Using EORTC QLQ-C30 assessment | Every 2 cycles for up to 24 months (each cycle is 28 days)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, EORTC QLQ-C30). All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Plasma Concentration of BR101801 (Bosmolisib) | Cycle 2 Day 1 and Day 1 of Cycle 3 (each cycle is 28 days)
  Blood samples were taken for the analyses of BR101801 in plasma at designated time points.
Adverse events | Approximately 24 months after a consent to the participation

IPD SHARING:
Plan to Share IPD: No